CLINICAL TRIAL: NCT01710020
Title: Phase 1, Open-Label Study Of The Pharmacokinetics, Non-Renal Clearance And Dialyzability Of CP-690,550 In Subjects With End-Stage Renal Disease Undergoing Hemodialysis
Brief Title: Pharmacokinetics And Dialysability Of CP-690,550 In Subjects With End-Stage Renal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A3921004
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-11

CONDITIONS: End-Stage Renal Disease; Hemodialysis
Keywords: CP-690; 550; pharmacokinetics; end-stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CP-690,550 (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — CP-690,550 10 mg oral powder for constitution

SUMMARY:
There were 2 study periods in this study. In the Period 1, CP-690,550 was to be administered approximately 1 to 2 hours following hemodialysis. If significant non-renal clearance of the drug occurred such that dialyzability of CP-690,550 could not be assessed in Period 1, a second period (Period 2) will be conducted. In Period 2, a single dose of drug will be administered approximately 4 hours prior to hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with end-stage renal disease
* Subjects need hemodialysis 3 times weekly

Exclusion Criteria:

* Subjects with evidence or history of clinically significant disease, excluding those common for subjects with End-Stage Renal Disease (ESRD).
* Subjects with any condition possibly affecting drug absorption.
* Subjects with malignancies with the exception of adequately treated basal cell carcinoma of the skin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-02; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Minneapolis, Minnesota

REFERENCES:
- [Derived] Krishnaswami S, Chow V, Boy M, Wang C, Chan G. Pharmacokinetics of tofacitinib, a janus kinase inhibitor, in patients with impaired renal function and end-stage renal disease. J Clin Pharmacol. 2014 Jan;54(1):46-52. doi: 10.1002/jcph.178. Epub 2013 Sep 30. PMID 24030917
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921004&StudyName=Pharmacokinetics%20And%20Dialysability%20Of%20CP-690%2C550%20In%20Subjects%20With%20End-Stage%20Renal%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 (10 mg OPC): Single oral dose of CP-690,550 10 milligram (mg) oral powder for constitution (OPC) 1 to 2 hours (hrs) post-hemodialysis in Period 1 followed by single oral dose of CP-690,550 10 mg OPC approximately 4 hours prior to hemodialysis in Period 2. A washout period of at least 14 days was maintained between each intervention period.
Period: Period 1
Arm/Group | CP-690,550 (10 mg OPC)
Started | 12
Completed | 11
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Washout Period (at Least 14 Days)
Arm/Group | CP-690,550 (10 mg OPC)
Started | 11
Completed | 11
Not Completed | 0
Period: Period 2
Arm/Group | CP-690,550 (10 mg OPC)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants enrolled in the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 45.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12, 16, 24 hours (hrs) post-dose in Period 1
Population: Analysis set included all participants who received study medication.
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Groups:
- CP-690,550 (Period 1): Single oral dose of CP-690,550 10 mg OPC 1 to 2 hours post-hemodialysis in Period 1.
Arm/Group | CP-690,550 (Period 1)
Number analyzed (Participants) | 12
nanogram*hour/milliliter (ng*hr/mL) | 396 (158)

2. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12, 16, 24 hrs post-dose in Period 1
Population: Analysis set included all participants who received study medication.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CP-690,550 (Period 1)
Number analyzed (Participants) | 12
ng*hr/mL | 385 (151)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12, 16, 24 hrs post-dose in Period 1
Population: Analysis set included all participants who received study medication.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | CP-690,550 (Period 1)
Number analyzed (Participants) | 12
nanogram/milliliter (ng/mL) | 106 (23.9)

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12, 16, 24 hrs post-dose in Period 1
Population: Analysis set included all participants who received study medication.
Measure: Median (Full Range); unit: hr
Arm/Group | CP-690,550 (Period 1)
Number analyzed (Participants) | 12
hr | 0.5 [0.5 to 0.5]

5. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12, 16, 24 hrs post-dose in Period 1
Population: Analysis set included all participants who received study medication.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | CP-690,550 (Period 1)
Number analyzed (Participants) | 12
hr | 3.46 (1.18)

6. Primary Outcome: Oral Clearance (CLpo)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. It was calculated by dividing given dose of drug with AUC.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 8, 12, 16, 24 hrs post-dose in Period 1
Population: Analysis set included all participants who received study medication.
Measure: Mean (Standard Deviation); unit: milliliter/minute (mL/min)
Arm/Group | CP-690,550 (Period 1)
Number analyzed (Participants) | 12
milliliter/minute (mL/min) | 501 (243)

7. Primary Outcome: Dialyser Clearance (CL HD) From 0 to 1 Hour
Description: Dialyser clearance was calculated as amount of drug in dialysate collected over a period of time (AHD) divided (/) by the product of fraction unbound of drug in plasma (fu), corresponding mid-time plasma concentration of drug (Cmid), and duration of dialysate collection period (tm). CL HD = AHD/(fu*Cmid*tm).
Time Frame: 0 to 1 hrs during hemodialysis started 4 hrs post-dose in Period 2
Population: Analysis set included all participants who received study medication. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mL/min
Groups:
- CP-690,550 (Period 2): Single oral dose of CP-690,550 10 mg OPC approximately 4 hours prior to hemodialysis in Period 2.
Arm/Group | CP-690,550 (Period 2)
Number analyzed (Participants) | 11
mL/min | 311 (124)

8. Primary Outcome: Dialyser Clearance (CL HD) From 1 to 2 Hour
Description: Dialyser clearance was calculated as amount of drug in dialysate collected over a period of time (AHD) divided by the product of fraction unbound of drug in plasma (fu), corresponding mid-time plasma concentration of drug (Cmid), and duration of dialysate collection period (tm). CL HD = AHD/(fu*Cmid*tm).
Time Frame: 1 to 2 hrs during hemodialysis started 4 hrs post-dose in Period 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CP-690,550 (Period 2)
Number analyzed (Participants) | 11
mL/min | 325 (138)

9. Primary Outcome: Dialyser Clearance (CL HD) From 2 to 3 Hour
Description: as for outcome 8
Time Frame: 2 to 3 hrs during hemodialysis started 4 hrs post-dose in Period 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CP-690,550 (Period 2)
Number analyzed (Participants) | 10
mL/min | 332 (135)

10. Primary Outcome: Dialyser Clearance (CL HD) From 3 to 4 Hour
Description: as for outcome 8
Time Frame: 3 to 4 hrs during hemodialysis started 4 hrs post-dose in Period 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CP-690,550 (Period 2)
Number analyzed (Participants) | 7
mL/min | 292 (111)

11. Secondary Outcome: Fraction of Unbound Drug (fu)
Description: Fraction of unbound drug (fu) is defined as the ratio of unbound drug concentration to the total drug concentration.
Time Frame: 2 hours post-dose in Period 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CP-690,550 (Period 1)
Number analyzed (Participants) | 11
ratio | 0.390 (0.042)

12. Other Pre Specified Outcome: Overall Dialyser Clearance (CL HD)
Description: as for outcome 8
Time Frame: 0 to 4 hrs during hemodialysis started 4 hrs post-dose in Period 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CP-690,550 (Period 2)
Number analyzed (Participants) | 11
mL/min | 318 (132)

13. Other Pre Specified Outcome: Dialyser Clearance (CL HD) From 3 to 3.5 Hour
Description: as for outcome 8
Time Frame: 3 to 3.5 hrs during hemodialysis started 4 hrs post-dose in Period 2
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CP-690,550 (Period 2)
Number analyzed (Participants) | 2
mL/min | 377 (200)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 (Period 1) | CP-690,550 (Period 2)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 5/12 | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 (Period 1) (N=12) | CP-690,550 (Period 2) (N=11)
Headache (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Ecchymosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 1
Cough increased (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.